CLINICAL TRIAL: NCT01928316
Title: Bioequivalence Study of Home-made and Imported Mizolastine Tablets in Healthy Volunteers
Brief Title: A Bioequivalence Study of Domestic (Made in China) and Imported Mizolastine Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017872; MIZOALY1001 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2013-08-19; First posted 2013-08-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Healthy; Bioequivalence; Mizolastine; Domestic; Imported
MeSH Terms: interventions — mizolastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental): Healthy male volunteers will receive single oral dose of 10 mg imported mizolastine tablet on Day 1 and single oral dose of 10 mg domestic (made in China) mizolastine tablet on Day 8.
  Interventions: Drug: Mizolastine domestic (made in China); Drug: Mizolastine (imported)
- Sequence B (Experimental): Healthy male volunteers will receive single oral dose of 10 mg domestic (made in China) mizolastine tablet on Day 1 and single oral dose of 10 mg imported mizolastine tablet on Day 8.
  Interventions: Drug: Mizolastine domestic (made in China); Drug: Mizolastine (imported)

INTERVENTIONS:
Drug: Mizolastine domestic (made in China) — Healthy male volunteers will receive 10 mg domestic (made in China) mizolastine tablets on Day 1 and Day 8
Drug: Mizolastine (imported) — Healthy male volunteers will receive 10 mg imported mizolastine tablets on Day 1 and Day 8

SUMMARY:
The purpose of the study is to evaluate the bioequivalence (the way in which different forms of the same drug are absorbed in the body) of single-dose administration of domestic (made in China) mizolastine tablets and imported mizolastine tablets given at the same dose in healthy volunteers

DETAILED DESCRIPTION:
This is a single-center, open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), crossover (method used to switch patients from one treatment arm to another in a clinical study) study. Approximately, 24 healthy volunteers will be enrolled in the study. Eligible volunteers will be randomly allocated to either Sequence A group or Sequence B group. On Day 1, volunteers from Sequence A group will receive imported mizolastine tablets and volunteers from Sequence B group will receive domestic mizolastine tablets. There will be a washout period (no treatment) of 7 Days. On Day 8, the two sequence groups will be switched. Volunteers from Sequence A group will receive domestic mizolastine and volunteers from Sequence B group will receive imported mizolastine tablets. Safety evaluations will include assessments of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination, which will be measured throughout the study. The maximum study duration for each volunteer will be approximately 16 days.

ELIGIBILITY:
Inclusion Criteria:

* No history of smoking
* Body mass index between 18 and 28 kilogram per square meter
* Health status considered good by the investigator according to physical examination, medical history, vital signs, electrocardiogram and clinical laboratory results
* Must be able to read and understand the informed consent form and sign the informed consent form before carrying out any operation related to the study

Exclusion Criteria:

* Health examination does not comply with the inclusion criteria
* Serious alcohol abuse
* Known allergy to active ingredients or excipients
* Habitual use of any drug including Chinese medicine

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Mizolastine (imported): Maximum Observed Plasma Concentration (Cmax) | Days 1, 2, 8, and 9 (Pre dose and Post dose 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 28, 36, 48 and 60 hours)
  The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration.
Mizolastine (domestic [made in China]): Maximum Observed Plasma Concentration (Cmax) | Days 1, 2, 8, and 9 (Pre dose and Post dose 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 28, 36, 48 and 60 hours)
  The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration.
Mizolastine (imported): Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Days 1, 2, 8, and 9 (Pre dose and Post dose 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 28, 36, 48 and 60 hours)
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Mizolastine (domestic [made in China]): Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Days 1, 2, 8, and 9 (Pre dose and Post dose 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 28, 36, 48 and 60 hours)
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Mizolastine (imported): Time to Reach Maximum Observed Plasma Concentration (Tmax) | Days 1, 2, 8, and 9 (Pre dose and Post dose 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 28, 36, 48 and 60 hours)
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Mizolastine (domestic [made in China]): Time to Reach Maximum Observed Plasma Concentration (Tmax) | Days 1, 2, 8, and 9 (Pre dose and Post dose 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 28, 36, 48 and 60 hours)
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.

SECONDARY OUTCOMES:
Number of volunteers with adverse events as a measure of safety and tolerability | Up to Day 16

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.